CLINICAL TRIAL: NCT00723645
Title: Rate and Predictors of Relapse in the Treatment of Hepatitis C in Real-life Clinical Practice in Spanish Hospitals (FAST-4)
Brief Title: Rate and Predictors of Relapse in the Treatment of Hepatitis C (Study P05181)
Acronym: FAST-4
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P05181
Record Dates: First submitted 2008-07-25; First posted 2008-07-29 (Estimated); Results first posted 2012-04-23 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2015-11

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PEG IFN alfa-2b + RBV: Adult participants with chronic hepatitis C who were treated for the first time with pegylated interferon alfa-2b plus ribavirin and achieved end-of-treatment response prior to the study. Participants received no treatment during this study.

SUMMARY:
This is an observational, multicenter, nationwide study where information will be collected on the follow-up of participants with chronic hepatitis C virus (HCV) who have a viral response at the end of treatment with pegylated interferon alfa-2b (PEG IFN alfa-2b) plus ribavirin (RBV) administered according to the directions on the products' labeling. No administration of treatment is planned as a result of study enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Participants with chronic hepatitis C virus (HCV)[any genotype] who received pegylated interferon alfa-2b plus ribavirin as first treatment for hepatitis C.
* Negative HCV RNA at the end of treatment (24 or 48 weeks according to the product labeling as appropriate), measured by the assay used at each institution. Only institutions using an assay with a limit of detection of 50 IU/mL or less will be eligible.

Exclusion Criteria:

* Women of childbearing potential (i.e., premenopausal women and women who are less than 6 months postmenopausal) who will not use an appropriate contraceptive method during the course of the clinical study. Appropriate contraceptives include double barrier methods (eg, diaphragm or condom plus spermicide), intrauterine device, oral, injectable or subcutaneous hormonal contraceptive, or surgically sterilized partner.
* Completed treatment with pegylated interferon alfa-2b plus ribavirin more than 4 weeks before study entry.
* Positive HCV RNA at the end of treatment (24 or 48 weeks according to the product labeling as appropriate).
* Participants treated for a period shorter than the enrollment period.
* Co-infection with Human Immumodeficiency Virus (HIV).
* Co-infected with Hepatitis B Virus (HBV).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects with chronic hepatitis C who were treated for the first time with pegylated interferon alfa-2b plus ribavirin and achieved end-of-treatment response.
Sampling Method: Non-Probability Sample
Enrollment: 279 (Actual)
Dates: Start 2008-04; Primary Completion 2010-04 (Actual); Study Completion 2011-02 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who had achieved a viral response prior to this study (negative for Hepatitis C Virus [HCV] ribonucleic acid [RNA] at the end of treatment as per product label) were recruited for follow-up on the present study.
Pre-assignment Details: A total of 279 participants enrolled in the study. Twenty-one participants failed screening and 258 participants were evaluable at Visit 1 (V1), which could be performed up to Week (Wk) 4 after the end of treatment.
Groups:
- PEG IFN Alfa-2b + RBV: Adult participants with chronic hepatitis C virus (HCV) who were treated for the first time with pegylated interferon alfa-2b plus ribavirin and achieved end-of-treatment response prior to the study. Participants received no treatment on this study.
Period: Visit 1 (≤4 Weeks Post-treatment)
Arm/Group | PEG IFN Alfa-2b + RBV
Started | 258
Completed | 258
Not Completed | 0
Period: Visit 2 (Week 24 Post-treatment)
Arm/Group | PEG IFN Alfa-2b + RBV
Started | 248 (10 discontinued before Visit 2; 7 lost to follow-up and 3 were HCV RNA+ before Wk 24)
Completed | 248
Not Completed | 0
Period: Visit 3 (Week 72 Post-treatment)
Arm/Group | PEG IFN Alfa-2b + RBV
Started | 187 (61 discontinued before V3; 26 lost to followup, 34 HCV RNA+ at Wk 24,1 death,1 HCV RNA not available)
Completed | 187
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | PEG IFN Alfa-2b + RBV
Number analyzed (Participants) | 258
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.72 (9.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 106
  Male | 152

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Relapse At 24 Weeks After the End Of Treatment (EOT)
Description: Relapse rate is defined as the percentage of participants with negative viral load (HCV RNA-) at EOT who have positive viral load (HCV RNA+) at 6 months after EOT.
  RNA= Ribonucleic Acid
Time Frame: From enrollment (≤4 weeks after end of treatment) to Week 24 post-treatment
Population: The evaluable population consisted of all enrolled participants who were virus negative at the end of treatment. 249 participants were evaluable for Week 24 (Visit 2).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | PEG IFN Alfa-2b + RBV
Number analyzed (Participants) | 249
Percentage of participants | 13.65 [9.39 to 17.92]

2. Secondary Outcome: Percentage of Participants Who Relapsed After EOT at Week 72 (Late Relapser)
Description: Late relapse was defined as having a Sustained Viral Response (SVR) at 24 weeks of follow-up and subsequently having a positive viral load 48 weeks later at Week 72.
  SVR was defined as negative for HCV RNA at Week 24 of follow-up.
Time Frame: From 24 weeks post-treatment to 72 weeks post-treatment
Population: The evaluable population consisted of all enrolled participants who were virus negative at the end of treatment and also virus-negative at Week 24 (Visit 2).
  187 participants completed Visit 2, 14 participants were excluded from analysis, and 173 participants were evaluable for Week 72 (Visit 3).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | PEG IFN Alfa-2b + RBV
Number analyzed (Participants) | 173
Percentage of participants | 0.58 [0 to 1.71]

ADVERSE EVENTS:
Arm/Group | PEG IFN Alfa-2b + RBV
Serious Adverse Events (participants affected / at risk) | 5/258
Other Adverse Events (participants affected / at risk) | 26/258
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PEG IFN Alfa-2b + RBV (N=258)
Drowning (General disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Spinal Hematoma (Nervous system disorders) | 1 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Schizophrenia, Paranoid Type (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PEG IFN Alfa-2b + RBV (N=258)
Anemia (Blood and lymphatic system disorders) | 13 (13)
Asthenia (General disorders) | 16 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No